CLINICAL TRIAL: NCT07223151
Title: Trading Sugar for Sparkles in Adolescents, A Sensory Approach for Reducing Added Sugar From Sweetened Beverages
Brief Title: A Sensory Strategy to Cut Sugary Beverages in African/American and Latine Adolescents
Acronym: SPARKLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nana Gletsu Miller (Other)
Collaborators: Purdue University (Other)
Responsible Party: Sponsor-Investigator, Nana Gletsu Miller, Associate Professor, Applied Health Science, Indiana University Bloomington, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB#25860; IRB#25860 (Other: Heartland Children's Nutrition Collaborative, supported by Riley Children's Foundation)
Record Dates: First submitted 2025-07-30; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Obesity, Adolescent; Dietary Sugars; Taste Perception; Insulin Resistance; Feeding Behavior
Keywords: Obesity; Adolescent; Sugar-Sweetened Beverages; Taste Perception; Insulin Resistance; Sweet Taste Preference; Latine Youth; African American Youth; Dietary Intervention; Beverage Replacement; Sugar Reduction; Sensory Evaluation; Randomized Controlled Trial
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Feeding Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three parallel intervention arms for 4 weeks: (1) replacement of sugary sodas with unsweetened, flavored sparkling water (USW), (2) replacement with sodas containing progressively reduced sugar levels (PRS), or (3) replacement with plain water (PW). All participants are followed for an additional 4-week period to assess maintenance of changes.
Masking Description: Not applicable. This is an open-label study; no parties are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unsweetened Sparkling Water (USW) (Experimental): Participants in this group will replace all sugar-sweetened sodas with flavored, unsweetened sparkling waters for 4 weeks.
  Interventions: Behavioral: Unsweetened Sparkling Water Replacement
- Progressively Reduced Sugar (PRS) (Experimental): Participants in this group will replace sugar-sweetened sodas with carbonated beverages that contain decreasing levels of sugar each week over a 4-week period, ending with a fully unsweetened sparkling water.
  Interventions: Behavioral: Progressively Reduced Sugar Beverage Replacement
- Plain Water (PW) (Active Comparator): Participants in this group will replace all sugar-sweetened sodas with plain, still water for 4 weeks. This arm serves as a control to compare outcomes against both the unsweetened sparkling water and gradually reduced sugar beverage interventions.
  Interventions: Behavioral: Plain Water Replacement

INTERVENTIONS:
Behavioral: Unsweetened Sparkling Water Replacement — Participants replace all sugar-sweetened sodas with flavored, unsweetened sparkling waters for 4 weeks.
  Arms: Unsweetened Sparkling Water (USW)
Behavioral: Progressively Reduced Sugar Beverage Replacement — Participants replace sugary sodas with beverages containing gradually decreasing sugar concentrations (weekly), ending with unsweetened sparkling water.
  Arms: Progressively Reduced Sugar (PRS)
Behavioral: Plain Water Replacement — Participants replace all sugar-sweetened sodas with plain, still water for 4 weeks. This serves as a comparator to evaluate sensory and metabolic changes.
  Arms: Plain Water (PW)

SUMMARY:
The goal of this clinical trial is to test whether replacing sugary sodas with unsweetened, flavored sparkling waters can reduce added sugar intake and improve health in Black/African American and Latine adolescents with obesity who prefer sweet-tasting beverages. The main questions it aims to answer are:

* Does replacing sugary sodas with water change liking for sugary drinks, and water?
* Do shifts in liking for sweetness lead to improved diet quality and cardiometabolic health?

Researchers will compare replacing sugary sodas with one of three alternative beverages: unsweetened sparkling water, plain water, and beverages with gradually reduced sugar to determine which strategy is most effective.

Participants will:

* Replace sugary sodas with study drinks for 4 weeks
* Complete taste tests to measure their liking for and sensory experience of sweetness over 8-weeks
* Provide dietary recalls, body measurements, and blood samples over 8-weeks

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effects of replacing sugar-sweetened sodas with unsweetened, flavored sparkling waters, progressively sugar-reduced sodas, or plain water in adolescents who are classified as "sweet-likers"-individuals who prefer higher concentrations of sugar in beverages. The study focuses on a high-risk group: adolescents ages 12-18 who self-identify as Black/African American or Latine and have obesity (BMI >95th percentile).

63 adolescents who are classified as sweet-likers and meet additional inclusion criteria will be enrolled in a randomized 3-arm intervention for 4 weeks, with an additional 4-week follow-up period. Participants will be randomized into one of the following groups:

USW (Unsweetened Sparkling Water): Replaces sodas with flavored, unsweetened carbonated water.

PRS (Progressively Reduced Sugar): Replaces sodas with carbonated beverages with decreasing sugar concentrations, ending with unsweetened carbonated water.

PW (Plain Water - Control): Replaces sodas with still, plain water.

Participants will replace all typical sugary sodas with study beverages during the 4-week intervention. Study assessments include sensory testing for liking, sweetness intensity, and "just about right" level of sweetness in sparkling and plain water at baseline, week 2, week 4, and week 8. Additionally, dietary intake (via 24-hour dietary recalls), anthropometrics (height, weight, waist circumference), blood pressure, and blood biomarkers (fasting glucose, insulin, triglycerides) will be measured at baseline, week 4, and week 8.

The primary hypothesis is that exposure to unsweetened beverages (especially in the USW and PRS groups) will reduce participants' liking for higher concentrations of sugar in beverages and increasing liking for lower concentrations of sugar in beverages. It is also hypothesized that these changes may correspond with improvements in cardiometabolic markers, particularly serum triglycerides. Insulin resistance (HOMA-IR), blood pressure, and body weight will also be measured but are less likely to shift in the relatively short time period (8 weeks).

This trial addresses the persistent challenge of high SSB consumption in racial and ethnic minority adolescents-a group that faces disproportionate risk of obesity, prediabetes, and cardiometabolic disease. By integrating sensory science with behavior change, this intervention seeks to develop more effective strategies to support reduced sugar intake in adolescents who have strong preferences for sweetness.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 12 to 18 who display a "sweet-liker" pattern, characterized by a preference for higher concentrations of sugar in beverages, specifically identifying 0.3M (10.3% sucrose) or above as their most liked sample.
* Have obesity (body mass index [BMI] > 95%). During screening, subjects' height and weight will be measured to calculate BMI, and BMI will be balanced across study arms using stratified randomization.
* Adolescents must also indicate a willingness to drink study beverages; not currently dieting/changing diet.

Exclusion Criteria:

* For the primary objective. Exclusion Criteria:

  * Adolescent participant is pregnant, since pregnancy affects taste perception
  * Participant is allergic or intolerant to the items we are testing.

For the secondary objective. Exclusion Criteria:

* Adolescent with type 1 or type 2 diabetes (self-declared or detected at screening visit through fasting glucose)
* Currently consume unsweetened, sparkling water two or more times per week.
* Adolescent participant is pregnant, since pregnancy affects taste perception
* Participant is allergic or intolerant to the items we are testing.
* Allergic or intolerant to the items that we are testing.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Liking ratings changes for sugar concentrations over time | Baseline, Week 2, Week 4, Week 8
  Our primary outcome is the interaction of time with liking for different sugar concentrations. We expect to observe a significant Time*Sugar Concentration interaction effect for these liking ratings. We expect the interaction term to show that higher concentrations of sugar had lower liking ratings by weeks 4 and 8 (compared to baseline), but that lower concentrations of sugar had higher liking ratings by weeks 4 and 8.
  Liking ratings are collected on a scale from -110 to 110, with internal markings at -100 Worst ever, -50 Dislike, 0 Neutral, 50 Like, 100 Best ever.

SECONDARY OUTCOMES:
Diet quality changes over time | Baseline, Week 4, Week 8
  We will use the ASA24 method to gather data on food intake. We will apply the Healthy Eating Index method to calculate diet quality. We expect to see improvements in diet quality at weeks 4 and 8 compared to baseline.
Serum triglyceride changes over time | Baseline, Week 4, Week 8
  A secondary outcome is the main effect of time on serum triglycerides. We expect to observe significant decreases in serum triglycerides at weeks 4 and 8 compared to baseline.
Change in fasting glucose over time | Baseline, Week 4, Week 8
  We will also evaluate fasting glucose by serum analysis.
Change in insulin resistance over time | Baseline, Week 4, Week 8
  We will also evaluate insulin resistance (HOMA-IR), which is a measure of fasting glucose multiplied by fasting insulin.
Change in BMI (body mass index) z-score | Baseline, Week 4, Week 8
  We will also evaluate BMI z-score for changes over time
Beverage Consumption Compliance | Baseline, Week 4, Week 8
  Participants report their beverage consumption and compliance will be assessed.
Change in Systolic Blood Pressure | Baseline, Week 4, Week 8
  Systolic Blood Pressure change over time will be evaluated.
Change in Diastolic Blood Pressure | Baseline, Week 4, Week 8
  Diastolic Blood Pressure change over time will be evaluated.
Change in Waist Circumference | Baseline, Week 4, Week 8
  Waist circumference will be evaluated over time.
Number of Participants experiencing tooth sensitivity or gastrointestinal symptoms | Week 4

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indiana University School of Public Health - Bloomington, Bloomington, Indiana
  - Indiana University Hospital, Indianapolis, Indiana
  - Purdue University, West Lafayette, Indiana

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the data collected from a minor population (adolescents), limited consent for data sharing. Future data sharing may be reconsidered following additional ethical review and participant re-consent where appropriate.

REFERENCES:
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Background] Wang J, Light K, Henderson M, O'Loughlin J, Mathieu ME, Paradis G, Gray-Donald K. Consumption of added sugars from liquid but not solid sources predicts impaired glucose homeostasis and insulin resistance among youth at risk of obesity. J Nutr. 2014 Jan;144(1):81-6. doi: 10.3945/jn.113.182519. Epub 2013 Nov 6. PMID 24198307
- [Background] Boushey CJ, Kerr DA, Wright J, Lutes KD, Ebert DS, Delp EJ. Use of technology in children's dietary assessment. Eur J Clin Nutr. 2009 Feb;63 Suppl 1(Suppl 1):S50-7. doi: 10.1038/ejcn.2008.65. PMID 19190645
- [Background] Bailey RL, Fulgoni VL, Cowan AE, Gaine PC. Sources of Added Sugars in Young Children, Adolescents, and Adults with Low and High Intakes of Added Sugars. Nutrients. 2018 Jan 17;10(1):102. doi: 10.3390/nu10010102. PMID 29342109
- [Background] Reedy J, Krebs-Smith SM. Dietary sources of energy, solid fats, and added sugars among children and adolescents in the United States. J Am Diet Assoc. 2010 Oct;110(10):1477-84. doi: 10.1016/j.jada.2010.07.010. PMID 20869486
- [Background] Banfield EC, Liu Y, Davis JS, Chang S, Frazier-Wood AC. Poor Adherence to US Dietary Guidelines for Children and Adolescents in the National Health and Nutrition Examination Survey Population. J Acad Nutr Diet. 2016 Jan;116(1):21-27. doi: 10.1016/j.jand.2015.08.010. Epub 2015 Sep 26. PMID 26391469
- [Background] Andes LJ, Cheng YJ, Rolka DB, Gregg EW, Imperatore G. Prevalence of Prediabetes Among Adolescents and Young Adults in the United States, 2005-2016. JAMA Pediatr. 2020 Feb 1;174(2):e194498. doi: 10.1001/jamapediatrics.2019.4498. Epub 2020 Feb 3. PMID 31790544
- [Background] Valicente V, Gletsu-Miller N, Running CA. Secondary Analysis of Sweetness Liking from Pilot Study Replacing Sugar Sweetened Soda with Flavored, Unsweetened Sparkling Water. J Am Nutr Assoc. 2025 Jan;44(1):1-13. doi: 10.1080/27697061.2024.2369819. Epub 2024 Jul 22. PMID 39037472
- See also: All IN for Health Research Studies - Study Listing for "Trading Sugar for Sparkles" — https://research-studies.allinforhealth.info/BFTI/